CLINICAL TRIAL: NCT05549531
Title: A Single-center, Open-label, Fixed-sequence Study to Investigate the Effect of Multiple-dose Itraconazole on the Pharmacokinetics of a Single Dose of 10 mg ACT-1004-1239 in Healthy Male Subjects
Brief Title: A Study to Investigate the Effect of Itraconazole on the Way the Body Absorbs, Distributes, and Gets Rid of ACT-1004-1239 Given as a Single Dose of 10 mg to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-086-103
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-1004-1239; Itraconazole

STUDY DESIGN:
Intervention Model Description: Open-label, fixed-sequence, drug-drug interaction (DDI) study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational and interaction treatment (Experimental): ACT-1004-1239 (10 mg) will be administered on Day 1 (in Treatment A) and Day 9 (in Treatment B2).
  Itraconazole (200 mg, o.d.) will be administered from Day 6 until Day 13. On Day 9, itraconazole will be administered concomitantly with ACT-1004-1239.
  Interventions: Drug: ACT-1004-1239 (10 mg); Drug: Itraconazole (200 mg, o.d.)

INTERVENTIONS:
Drug: ACT-1004-1239 (10 mg) — ACT-1004-1239 will be administered as 1 capsule of 10 mg strength to be taken under fed conditions.
Drug: Itraconazole (200 mg, o.d.) — Itraconazole 200 mg will be administered as capsules (2 x 100 mg capsule) to be taken under fed conditions.

SUMMARY:
A study to investigate the effect of itraconazole on the way the body absorbs, distributes, and gets rid of ACT-1004-1239 given as a single dose of 10 mg to healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male subject aged between 18 and 55 years (inclusive) at Screening.
* Negative SARS-CoV-2 test or valid EU Digital COVID-19 Recovery Certificate prior to Day -1.
* A male subject with a partner of childbearing potential must use adequate contraception (i.e., condom) from first study treatment administration up to at least 30 days after EOS or premature study discontinuation (i.e., safety follow-up).

Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Participation in a clinical study involving study treatment administration within 12 weeks prior to Screening or in more than 2 clinical studies within 1 year prior to Screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
* Previous treatment with any prescribed medications (including vaccines such as COVID-19 vaccine) or OTC medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks prior to first study treatment administration.
* Positive results from urine drug and alcohol screen at Screening, on Day -1.
* Positive serology results for HIV1 and HIV2 antibodies, hepatitis B surface antigen, and hepatitis C antibodies at Screening.
* Any signs or symptoms of an acute clinically relevant illness within 4 weeks prior to Screening (e.g., bacterial, viral, or fungal infection) as judged by the investigator.
* Any cardiac condition or illness that may jeopardize the safety of the study subject as per the investigator's judgment based on medical history or 12-lead ECG measured at Screening.
* Any immunosuppressive treatment within 6 weeks or 5 x t½, whichever is longer, before first study treatment administration.
* Clinically relevant abnormalities or abnormalities of uncertain clinical significance on 12-lead ECG, measured after 5 min in a supine position at Screening or on Day -1.
* Baseline QTc interval >450 ms or <350 ms at Screening or on Day -1.
* Alanine aminotransferase, aspartate aminotransferase, or creatinine kinase values above the upper limit of the normal range at Screening.
* Estimated renal creatinine clearance (CrCL) below 90 mL/min, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average surface area of 1.73 m2 at Screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter for plasma ACT-1004-1239: Cmax | Blood samples for PK analysis will be taken prior to study treatment administration and at multiple timepoints from Day 1 to Day 6 (Treatment period A) and from Day 9 to Day 14 (Treatment period B2; total duration: 12 days).

SECONDARY OUTCOMES:
Pharmacokinetic parameters for plasma ACT-1004-1239: tmax | Blood samples for PK analysis will be taken prior to study treatment administration and at multiple timepoints from Day 1 to Day 6 (Treatment period A) and from Day 9 to Day 14 (Treatment period B2; total duration: 12 days).
Pharmacokinetic parameters for plasma ACT-1004-1239: AUC0-inf | Blood samples for PK analysis will be taken prior to study treatment administration and at multiple timepoints from Day 1 to Day 6 (Treatment period A) and from Day 9 to Day 14 (Treatment period B2; total duration: 12 days).
Pharmacokinetic parameters for plasma ACT-1004-1239: t1/2 | Blood samples for PK analysis will be taken prior to study treatment administration and at multiple timepoints from Day 1 to Day 6 (Treatment period A) and from Day 9 to Day 14 (Treatment period B2; total duration: 12 days).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- BlueClinical Phase 1, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huynh C, Dingemanse J, Meyer Zu Schwabedissen HE, Fonseca M, Sidharta PN. The effect of itraconazole, a strong CYP3A4 inhibitor, on the pharmacokinetics of the first-in-class ACKR3/CXCR7 antagonist, ACT-1004-1239. Clin Transl Sci. 2024 Jul;17(7):e13883. doi: 10.1111/cts.13883. PMID 39010703